CLINICAL TRIAL: NCT04842669
Title: Effects of Low Level Laser Therapy On Exercise Induced Muscle Damage in Wrist Flexors Of Untrained Young Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00864 Kirran Sikandar
Record Dates: First submitted 2021-04-10; First posted 2021-04-13 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Wrist Injuries
Keywords: exercise induced muscle damage; wrist flexor; low level laser therapy
MeSH Terms: conditions — Wrist Injuries | interventions — Low-Level Light Therapy; Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level laser therapy (Experimental): Low level laser therapy
  Interventions: Other: low level laser therapy
- Conservative treatment (Active Comparator): Conservative treatment
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Other: low level laser therapy — Endo-laser 422 with interchangeable laser probes will be used for the purpose. It is a 2-channel unit and is software operated. For treatment of small surfaces with mono laser there are diodes of 25, 100 and 500 milliWatt.Frequency will be adjusted to 500 Hz, dose 0.1/cm2 with time duration of 1-5 minutes.
  Arms: Low level laser therapy
Other: Conservative treatment — (Topical ibuprofen gel) for muscle soreness will be provided
  Arms: Conservative treatment

SUMMARY:
The main aim of the current study is to investigate the effects of Low-level Laser Therapy on exercise-induced muscle damage of wrist flexors in untrained young adults. A randomized controlled trial will be conducted at Sargodha Medical College, University of Sargodha. The sample size calculated is 16. The participants will be divided into two equal group; 1) Interventional group (Low level laser therapy), 2) Control group (conventional) each having 8 participants. The study duration will be six months after approval from Research board. Blocked randomization sampling technique will be used. The subjects will be randomly assigned to any of the interventional or control group. Interventional group will further be allocated to prophylactic or therapeutic group. Only Un-trained young Adults, Aged 19-25 (under-graduate/college and university students) without gender discrimination will be included in the study. Tools used in the study will be TALAG Scale (Soreness assessment), Goniometer (ROM), Algometer (Pressure¬-pain Threshold), Electronic digital hand Dynamometer (Grip Strength) and PRS (Perceived Recovery Status Scale). Data will be collected at baseline, 1hr, 24hr, 72hr, 96hr, 120hr, 148hr, 168hr and 192 hrs after the induction protocol.

DETAILED DESCRIPTION:
Wrist flexors play a crucial role in hand function. This group of small muscles is of high importance in our day to day tasks like carrying heavy objects and for activities in which forceful and/or rapid wrist flexions are required. Apart from this, the wrist flexors have a distinctive neural control as compared to the other surrounding musculature.

Muscle exhaustion that is induced after eccentric exercise, can either be of acute onset or delayed onset. Exercise induced muscle soreness that persists for about 4 to 6 hours before it returns to pre-exercise level is termed as acute soreness. On the other hand, muscle soreness beginning at 8 to 24 hours after eccentric exercise, with peak level at 24 to 48 hours is known as delayed soreness. Delayed-Onset Muscle Soreness (DOMS) is a common neuromuscular condition characterized by increased sensitivity to pain that is apparent with unaccustomed or vigorous exercise, a day after performance. DOMS becomes evident about 6-8 hours after an intense exercise bout and peaks at approximately 24-72 hours post-exercise. During first few hours of intensive exercise metabolism get disturbed that leads to inefficient physical activity and performance. Prolonged metabolic disturbances and physical activity and performance impairment progressing to days ultimately induce tissue damage that we call as delayed-onset muscle soreness. Event that produces muscle soreness is suggested as a mechanical disruption of sarcomeres leading to swelling of injured muscle fibers thus initiating an inflammatory response leading to the excitement of nociceptors.

Exercise-induced muscle injury is similar in pathological change and pathogenic mechanism in humans and animals. Human beings and animals have shown parallel reactions to changes caused by muscle damage induced by eccentric exercises. The beginning of initial exercise-induced muscle damage may be draining but is pain free. Later on, after 8-24 hours of muscle damage initiation, the subsequent inflammation results in delayed onset of muscle soreness.

It has been assumed that whenever an un-habitual physical exercise is carried out by a person then muscle injury occurs. A high level of muscle injury is associated with eccentric activities. Muscle injury is more likely to occur in untrained individuals who start practicing exercise. Furthermore, incidence of muscle injury is more common with exercises involving eccentric activities. Loss of strength, muscle inflammation, high level of muscle proteins in blood and delayed onset of muscle soreness DOMS are considered to be the expected outcomes of muscle injury. Different electro-physical modalities are being used by Physical therapists. In many conditions, improved healing and functioning are achieved by the use of these electro-physical modalities. Some animal studies have also reported the positive role of Low-Level Laser Therapy, when used in optimal parameters of irradiations, in enhancing the muscle healing and decreasing inflammation. Increased amount and activity of mitochondria and increased cross-sectional area of muscle fiber is associated with training. Increased muscle mass and improved mitochondrial function result in shift in muscle fiber type composition, from type two B to type Two A, and an increase in local glycogen storage capability. These combined adaptations make specialized athletes chiefly different from untrained people.

Several studies performed on human and animals evidenced the action of Low-level Laser Therapy in achieving therapeutic and physiological effects involving improvement of muscle functioning through interaction with biological tissues. Decrease in muscle fatigue has been reported by several researchers with the application of Laser Therapy before exercises that induces fatigue while considerable functional enhancement has also been evidenced by some investigators with Laser application after performing fatigue inducing exercises. Therapeutic effect of LLLT may be explained by mechanisms involving improved microcirculation of tissue, anti-inflammatory effect, decreased oxidative stress and decrease in tissue ischemia.

In 2016, a study was conducted to evaluate the effects of low level laser therapy on post exercise recovery of skeletal muscle and improvement in muscle performance and function. The conclusion of this study was that pre-exercise treatment with low level laser therapy increases muscle performance along with improvement in biochemical markers associated with inflammation and muscle injury.

In August 2011, Wouber Hérickson de Brito and fellows carried out a comparative study to investigate whether muscle performance could be increased with endurance training associated with LLLT when compared to the same training without LLLT. Results suggested a great decrease in fatigue when training was combined with LLLT, thus improving the muscle performance.

In August 2010, a study was carried out to find out the effectiveness of low-level laser therapy (LLLT) on muscle performance, fatigue development, and biochemical markers of post-exercise recovery on bicep muscle. Results clearly suggested that endurance for repetitive elbow flexion has been increased with the application of LLLT before exercise while levels of reactive protein, creatine kinase and blood lactate has been decreased after performance of exercise.

In July 2010, to investigate the effects of Low-level laser therapy before eccentric exercise on muscle damage markers in humans. It was concluded that LLLT therapy when given before performance of eccentric exercise, accelerated the increase of muscle proteins in the blood serum and the decrease in muscle force.

In July 2011, a study was carried out to compare the effects of Red (660 nm) and infrared (830 nm) low-level laser therapy in skeletal muscle fatigue in humans. The study showed that both red and infrared LLLT are effective in delaying the development skeletal muscle fatigue and in improvement of skeletal functioning.

In August 2009, to investigate the Effects of Low-Level Laser Irradiation on Skeletal Muscle Injury after Eccentric Exercise. It was the first study performed on animal model to investigate these effects. It was concluded that Low-level He-Ne laser therapy exerts therapeutic effects by improving anti-oxidative capacity of muscle as well as decreasing the inﬂammatory reaction.

ELIGIBILITY:
Inclusion Criteria:

* Un-trained young Adults

Exclusion Criteria:

* Any Trauma
* Any psychological condition
* Participation in any scheduled Physical training
* Athlete population
* Use of any nutritional supplement

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS): | 8th day (192 hours)
  The Numeric Rating Scale is an 11 point scale where the end points are the extremes of no pain and pain as bad as it could be, or worst pain. Numerical Rating Scale has good sensitivity and generates data that can be statistically analyzed for audit purposes.
  Measurements were done at 24, 48, 72, 96,120, 144 and 168, and 192 hours at the same time of the day.
TALAG Scale (Soreness assessment): | 8th day (192 hours)
  TALAG scale will be used to assess the perceived soreness. It consists of points 1-7 on scale. The minimum level 1 with no pain and a maximum point 7 with unbearably painful.Measurement of all dependent variables at 24, 48, 72, 96,120, 144 and 168, and 192 hours after eccentric exercise were taken at the same time of the day.
Goniometer | 8th day (192 hours)
  Physical therapists widely use goniometer for measurement of different joint ranges to evaluate any ROM limitation. The universal full circle goniometer is the preferred instrument for measuring ROM.Measurement of all dependent variables at 24, 48, 72, 96,120, 144 and 168, and 192 hours after eccentric exercise were taken at the same time of the day.
Pressure-pain Threshold by Algometer | 8th day (192 hours)
  Algometer is a reliable tool for measuring pressure pain threshold(22).The Pressure Pain Threshold will be evaluated using an analogue algometer (Baseline, 60 pounds capacity) by applying vertical pressure. To stimulate the participant's pain, the pressure will be increased at a rate of 1kg/cm2.Measurements will be taken pre and post treatment for 2 times during study. Measurement of all dependent variables at 24, 48, 72, 96,120, 144 and 168, and 192 hours after eccentric exercise were taken at the same time of the day.
Electronic digital hand Dynamometer | 8th day (192 hours)
  Grip strength will be evaluated with an electronic digital hand dynamometer as per recommendations. Measurement of all dependent variables at 24, 48, 72, 96,120, 144 and 168, and 192 hours after eccentric exercise were taken at the same time of the day.

SECONDARY OUTCOMES:
Perceived Recovery (Perceived Recovery Status Scale): | 8th day (192 hours)
  PRS scale is a convenient, noninvasive marker of recovery relative to subsequent training.
  This scale consist of 10 points from 0 -10 with the minimum value 0 for very poorly recovered and maximum 10 value for very well recovered.Measurement of all dependent variables at 24, 48, 72, 96,120, 144 and 168, and 192 hours after eccentric exercise were taken at the same time of the day.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Sargodha Medical College (University of Sargodha), Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No